CLINICAL TRIAL: NCT04980573
Title: The Effects of Aromatherapy on Post COVID-19 Fatigue: A Randomized, Double Blind, Controlled Trial
Brief Title: Essential Oils and Post COVID-19 Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Collaborators: Young Living Essential Oils (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-07-0300
Record Dates: First submitted 2021-07-26; First posted 2021-07-28 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Covid19; Fatigue
Keywords: essential oils; aromatherapy; energy
MeSH Terms: conditions — COVID-19; Fatigue | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive a bottle of plant-based oil to inhale twice daily for 14 days.
  Interventions: Other: Aromatherapy
- Placebo (Placebo Comparator): Participants receive a bottle of inert oil to inhale twice daily for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aromatherapy — The aromatherapy intervention consists of inhaling a fragrant oil extracted from citrus peels, plant resins, and leaves.
  Arms: Intervention
Other: Placebo — The placebo intervention consists of inhaling an oil extracted from inert plant matter.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of plant based aromas on energy levels among otherwise healthy female survivors of COVID-19.

DETAILED DESCRIPTION:
After being informed about the study, participants will provide informed consent, then will be randomized into one of two groups in a 1:1 ratio. Participants will either inhale an inert blend twice a day or an active aroma twice a day for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-49
* Lives in the United States
* Otherwise Healthy
* COVID-19 Diagnosis between December 1, 2020 and March 31, 2021
* Decreased energy or fatigue at a level that was not present prior to the diagnosis

Exclusion Criteria:

* Positive COVID-19 test any time before December 1, 2020
* Positive COVID-19 test any time after March 31, 2021
* COVID vaccine of any type scheduled during the intervention period or the week prior to the start of the study
* Allergy to any of the ingredients
* Pregnant, trying to conceive, or breastfeeding
* Regular smokers in the home
* Abnormal pulmonary function
* Chest pain
* Recurring headaches
* Uncontrolled hypertension
* Chronic Fatigue Syndrome diagnosis
* Persistent fatigue prior to COVID-19 diagnosis
* Hypothyroidism

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on self-representation of gender and is restricted to women.
Enrollment: 47 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Multidimensional Fatigue Symptom Inventory (MFSI) at day 14. | Baseline and Day 14
  The MFSI is a validated, 83 question scale measuring fatigue levels across ten domains. Each question is scored from 0-5 on a Likert scale, with higher scores indicating higher levels of fatigue.

SECONDARY OUTCOMES:
Change from baseline to day 14 on the Patient Health Questionnaire (PHQ-9) | Baseline and Day 14
  This survey includes 9 questions regarding levels of depression. Each question is scored from 0-3 on a Likert scale, with higher scores indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No